CLINICAL TRIAL: NCT01852331
Title: The Herbal Medicine Peony-Glycyrrhiza Decoction (PGD) as an Adjunctive Therapy to Treat Antipsychotic-induced Hyperprolactinemia in Patients With Schizophrenia: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Peony-Glycyrrhiza Decoction (PGD) for Antipsychotic-induced Hyperprolactinemia in Patients With Schizophrenia
Acronym: PGD-RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Kowloon Hospital, Hong Kong (Other); Queen Mary Hospital, Hong Kong (Other); Capital Medical University (Other); Xijing Hospital (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 11-274
Record Dates: First submitted 2013-05-06; First posted 2013-05-13 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia; Schizophrenic Disorder; Hyperprolactinemia; Hyperprolactinaemia
Keywords: Schizophrenia; Schizophrenic Disorder; Hyperprolactinemia; Hyperprolactinaemia; Chinese herbal medicine; Traditional Chinese medicine; Peony-Glycyrrhiza Decoction; PGD; Glycyrrhiza Radix; Liquorice Root; Gancao; Paeoniae Alba Radix; White Peony Root; Baishao
MeSH Terms: conditions — Schizophrenia; Hyperprolactinemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PGD granules (Active Comparator): While continuing current antipsychotic medications, subjects will receive adjunctive Peony-Glycyrrhiza Decoction (PGD) granules (equivalent to 45 g raw materials in total per day). They need to take the granules two times a day, each time one sachet (aluminum foil pack of 9g, tear open and empty contents into a cup, add 200ml hot water, stir until dissolute completely, and drink the preparation when warm), for a consecutive of 16 weeks.
  Interventions: Drug: PGD granules
- Placebo (Placebo Comparator): While continuing current antipsychotic medications, subjects will receive adjunctive treatment with placebo granules. They need to take the placebo granules two times a day, each time one sachet (aluminum foil pack of 9g, tear open and empty contents into a cup, add 200ml hot water, stir until dissolute completely, and drink the preparation when warm), for a consecutive of 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PGD granules — The preparation of Peony-Glycyrrhiza Decoction (PGD) granules is in compliance with Pharmacopoeia of the People's Republic of China and Good Manufacturing Practice (GMP). Briefly, sliced, broiled Paeoniae Alba Radix and Glycyrrhizae Radix in a ratio of 1:1 in weight will be immersed and boiled in an 8-fold volume of distilled water for 2.5 hours. This process will be repeated twice. The extract solution will be pooled and concentrated into granule form. Weight of the resulting granules contained in two 9g-sachet packs (to be taken in one day) is equivalent to 45 g raw herbal materials which are supplied for one day.
  Arms: PGD granules
Drug: Placebo — The placebo granules are prepared to be identical to PGD granules in smell, taste and color.
  Arms: Placebo

SUMMARY:
The investigators hypothesize that Peony-Glycyrrhiza Decoction (PGD) adjunctive therapy could reduce the incidence of prolactin (PRL)-related adverse events in patients with schizophrenia and suppress antipsychotic-induced elevation of PRL levels.

This is a placebo-controlled trial conducted in schizophrenic patients to determine whether PGD adjunctive treatment could produce greater biochemical and clinical improvement on hyperprolactinemia (hyperPRL) compared to placebo treatment.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness that affects 0.7-1.1% of the worldwide population. Most patients who develop a chronic course with frequent relapses and exacerbation of psychosis are required to have long-term treatment. The clinical outcomes of antipsychotic pharmacotherapy are limited, largely due to various adverse side effects. Hyperprolactinemia (hyperPRL) is the most challenging among them. Dopamine agonists may be used for hyperPRL if it does not improve after the reduction of antipsychotic doses. However, this may aggravate psychosis and abnormal involuntary movements, which may be a greater risk than hyperPRL itself.

Chinese herbal medicine called Peony-Glycyrrhiza Decoction (PGD) has been widely introduced into the treatment of various conditions associated with hyperPRL in China and Japan. In our series of in-vitro experience it was found that PGD can significantly suppress PRL concentration in the cultured medium in a dose-dependent manner. Our recent open-labelled pilot study demonstrated that PGD significantly suppressed risperidone-induced elevation of blood PRL levels and produced a greater improvement on hyperPRL-related symptoms compared to dopamine agonist bromocriptine. Empirical and experimental evidence also confirmed that PGD and its individual herbal preparations possess a high safety profile.

The encouraging results obtained from our laboratory and clinical pilot studies, together with findings of previous studies, have warranted an extensive controlled trial to further determine PGD as an effective therapy for the treatment of antipsychotic-induced hyperPRL.

ELIGIBILITY:
Inclusion Criteria:

* have a primary diagnosis of schizophrenia or schizoaffective disorder based on International Classification of Diseases (10th edition);
* under antipsychotic medications for at least three months and current conditions are stable, indicated by no difficulty to communicate with investigators and give informed consent;
* have developed at least one overt hyperPRL-associated symptom, including oligomenorrhoea (infrequent, irregularly timed episodes of bleeding occurring at intervals of more than 35 days from the previous menstrual cycle), amenorrhoea (the absence of menstruation for three menstrual cycles or 6 months), galactorrhea, decreased libido, anorgasmia or erectile dysfunction; and
* serum PRL levels are >24 ng/ml (or 1043.472 pmol/l) in female or >19 ng/ml (or 826.082 pmol/l) in male.

Exclusion Criteria:

* unstable medical conditions;
* suicidal ideas or attempts or aggressive behavior;
* history of alcoholism in the past one year, characterized by compulsive and uncontrolled consumption of alcohol, despite the realization of its negative effects on health, relationship, and social standing;
* history of drug abuse in past one year;
* currently treated with Chinese medicine or other natural products;
* allergic history of herbal medicine;
* pre-existing hyperPRL symptoms not associated with antipsychotic treatment; and
* pregnant and lactating women and those who refuse to use contraception during the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Positive and Negative Syndrome Scale (PANSS) at 8 weeks and 16 weeks | baseline, week 8 and week 16
  The severity of psychotic symptoms will be assessed using the Positive and Negative Syndrome Scale (PANSS)
Changes from baseline Clinical Global Impression (CGI) score at 8 weeks and 16 weeks | baseline, week 8 and week 16
  The severity of psychotic symptoms will be assessed using the Clinical Global Impression (CGI).
Changes from baseline Simpson-Angus Rating Scale (SAS) at 8 weeks and 16 weeks | baseline, week 8 and week 16
  The Simpson-Angus Rating Scale (SAS) will be used to evaluate antipsychotic-induced abnormal involuntary movement symptoms.
Changes from baseline Abnormal involuntary movement scale (AIMS) at 8 weeks and 16 weeks | baseline, week 8 and week 16
  The abnormal involuntary movement scale (AIMS) will be used to evaluate antipsychotic-induced abnormal involuntary movement symptoms.

SECONDARY OUTCOMES:
Change from baseline scores of Prolactin Related Adverse Event Questionnaire (PRAEQ) at 8 weeks and 16 weeks | baseline, week 8 and week 16
  Menstrual disturbances, breast symptoms and penile function will be assessed using the Prolactin Related Adverse Event Questionnaire (PRAEQ).
Change from baseline scores of Udvalg for Kliniske Undersøgelser Side Effect Rating Scale (UKU) at 8 weeks and 16 weeks | baseline, week 8 and week 16
  Other adverse effects will be assessed using the Udvalg for Kliniske Undersøgelser Side Effect Rating Scale (UKU).

OTHER OUTCOMES:
Changes from baseline serum prolactin levels at 8 weeks and 16 weeks | baseline, week 8 and week 16
  Serum concentrations of serum prolactin will be measured using chemiluminescent immunoassay (CLIA).
Changes from baseline serum estradiol levels at 8 weeks and 16 weeks | baseline, week 8 and week 16
  Serum concentrations of estradiol will be measured using chemiluminescent immunoassay (CLIA).
Changes from baseline serum testosterone levels at 8 weeks and 16 weeks | baseline, week 8 and week 16
  Serum concentrations of testosterone will be measured using chemiluminescent immunoassay (CLIA).

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin Zhang, MMed, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (4):
- China (4):
  - Xijing Hospital, Xian, Shanxi
  - Beijing Anding Hospital, Beijing
  - Department of Psychiatry, Queen Mary Hospital, Hong Kong
  - Department of Psychiatry, Kowloon Hospital, Kowloon

REFERENCES:
- [Derived] Man SC, Li XB, Wang HH, Yuan HN, Wang HN, Zhang RG, Tan QR, Wong HK, McAlonan GM, Wang CY, Zhang ZJ. Peony-Glycyrrhiza Decoction for Antipsychotic-Related Hyperprolactinemia in Women With Schizophrenia: A Randomized Controlled Trial. J Clin Psychopharmacol. 2016 Dec;36(6):572-579. doi: 10.1097/JCP.0000000000000607. PMID 27755159